CLINICAL TRIAL: NCT06765343
Title: Efficacy of Guided Biofilm Therapy in Pediatric Patient: a Randomized Clinical Trial
Brief Title: Efficacy of Guided Biofilm Therapy in Pediatric Patient
Acronym: BABYPLAK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Magda Mensi, Researcher, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BABYPLAK NP 5675
Record Dates: First submitted 2024-11-28; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Oral Hygiene, Oral Health; Pediatric Pain and Anxiety
Keywords: guided biofilm therapy; discloser agent; airflowing; polishing; patient feedback
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial, mono-centric, 2 by 2 parallel
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Guided biofilm therapy with plaque disclosing (GBT+) (Experimental): Participants assigned to the GBT+ receive professional air-flowing oral hygiene with erythritol powder followed by ultrasonic calculus removal, guided by a plaque disclosing agent. At the and of the treatment the investigator notes the treatment time, places the disclosing agent, takes a standardised intra-oral picture, records the FMPS (full mouth plaque score) and administers a feedback questionnaire to the participant.
  Interventions: Device: Plaque disclosing agent; Device: Guided Biofilm Therapy
- Guided biofilm therapy without plaque disclosing (GBT-) (Experimental): Participants assigned to the GBT+ receive professional air-flowing oral hygiene with erythritol powder followed by ultrasonic calculus removal, without the guide of a plaque disclosing agent. At the and of the treatment the investigator notes the treatment time, places the disclosing agent, takes a standardised intra-oral picture, records the FMPS (full mouth plaque score) and administers a feedback questionnaire to the participant.
  Interventions: Device: Guided Biofilm Therapy
- Ultrasonic debridement and polishing with plaque disclosing (US+C+) (Experimental): Participants assigned to the US+C+ receive traditional professional oral hygiene (ultrasonic tip followed by rubber cup and polishing paste) guided by a plaque disclosing agent. At the and of the treatment the investigator notes the treatment time, places the disclosing agent, takes a standardised intra-oral picture, records the FMPS (full mouth plaque score) and administers a feedback questionnaire to the participant.
  Interventions: Device: Plaque disclosing agent; Device: Ultrasonic debridement and polishing
- Ultrasonic debridement and polishing without plaque disclosing (US+C-) (Active Comparator): Participant assigned to the US+C- receive traditional professional oral hygiene (ultrasonic tip followed by rubber cup and polishing paste) without the guide of a plaque disclosing agent. At the and of the treatment the investigator notes the treatment time, places the disclosing agent, takes a standardised intra-oral picture, records the FMPS (full mouth plaque score) and administers a feedback questionnaire to the participant.
  Interventions: Device: Ultrasonic debridement and polishing

INTERVENTIONS:
Device: Plaque disclosing agent — Dye agent binding to oral biofilm and plaque for visual detection
  Arms: Guided biofilm therapy with plaque disclosing (GBT+); Ultrasonic debridement and polishing with plaque disclosing (US+C+)
Device: Guided Biofilm Therapy — Utilisation of a air-polishing device conveying a jet of air, water and erythritol powder for plaque debridement on dental surfaces, followed by calculus removal with an ultrasonic scaler
  Arms: Guided biofilm therapy with plaque disclosing (GBT+); Guided biofilm therapy without plaque disclosing (GBT-)
Device: Ultrasonic debridement and polishing — Removal of plaque and calculus with an ultrasonic scaler, followed by surface polishing with a rubber cup and abrasive paste
  Arms: Ultrasonic debridement and polishing with plaque disclosing (US+C+); Ultrasonic debridement and polishing without plaque disclosing (US+C-)

SUMMARY:
The present parallel randomized clinical trial aims to assess the efficacy of a plaque disclosing agent (PDA) and air-flowing with erythritol powder (Guided Biofilm Therapy) in the removal of biofilm and plaque in paediatric participants during professional oral hygiene, compared with ultrasonic debridement.

The participants will be divided in four groups and receive:

* Guided Biofilm Therapy with plaque disclosing agent (GBT+)
* Guided Biofilm Therapy without plaque disclosing agent (GBT-)
* Ultrasonic debridement and polishing with plaque disclosing agent (US+C+)
* Ultrasonic debridement and polishing without plaque disclosing agent (US+C-)

Clinical and image software analysis (ImageJ) of residual plaque will be performed.

DETAILED DESCRIPTION:
Oral biofilm is not easily detectable visually, so its removal can be difficult. Using a plaque disclosing agent to highlight biofilm and plaque could aid during its removal and may be beneficial.

In paediatric patients, often times it is more difficult to perform professional oral hygiene because of lack of compliance. Our hypothesis is that the visual guide of the plaque disclosing might help obtaining a better result in terms of plaque removal. Moreover, the use of air-flowing could lead to several advantages compared to traditional professional oral hygiene (ultrasonic debridement and polishing cups), such as increased comfort and compliance, shorter treatment time, easier access to difficult areas and the minimal-invasiveness on soft and hard tissue.

The study is a mono-centric, pragmatic, single-blinded, randomized clinical trial (RCT) of parallel design.

The primary outcome is the Residual Plaque Area (RPA) expressed in percentage of area with residual plaque highlighted by disclosing plaque agent. Secondary outcomes are Full Mouth Plaque Score (FMPS), treatment time and participants' feedback.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form (pediatric patient and parent).
* Male and female subjects, aged 6 -12 years, inclusive.
* Good general health (ASA I e II)
* With at least 80% of dentition present
* With at least 8/12 frontal dental elements.

Exclusion Criteria:

* Not willing to follow the agreed protocol.
* Presence of orthodontic appliances.
* Tumors or significant pathology of the soft or hard tissues of the oral cavity.
* Current radiotherapy or chemotherapy.
* History of allergy to Erythritol.
* History of adverse reactions to lactose or fermented milk products.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-09-12 (Actual)

PRIMARY OUTCOMES:
Residual Plaque Area (RPA) | Through study completion, an average of 1 year
  The percentage of area on which plaque is still present, as revealed by reapplication of a plaque disclosing agent, at the end of the treatment session. An intra-oral picture is taken and it is analyzed with a specific software: ImageJ

SECONDARY OUTCOMES:
Full Mouth Plaque Score (FMPS) | Through study completion, an average of 1 year
  The percentage of full mouth residual plaque detected with plaque disclosing agent after the treatment
Time Session | Through study completion, an average of 1 year
  The duration of treatment is noted and compared between groups
Participant Feedback | Through study completion, an average of 1 year
  A satisfaction questionnaire (VAS Scale) is administered to the participant
Operator Feedback | Through study completion, an average of 1 year
  A satisfaction questionnaire (VAS Scale) is administered to the operator

CONTACTS AND LOCATIONS:
Locations (1):
- ASST Spedali Civili di Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT06765343/Prot_SAP_000.pdf